CLINICAL TRIAL: NCT05822076
Title: Evaluation of Influence of Thoracic Paravertebral Block on Cardiac Repolarization
Brief Title: Influence of Thoracic Paravertebral Block on Cardiac Repolarization
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radosław Owczuk, Clinical Professor, Head of Department of Anesthesiology and Intensive Care, Medical University of Gdansk
Other Study IDs: NKBBN/948/2022
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Paravertebral Block; QT Interval
Keywords: QT Interval; Transmural dispersion of repolarization; Paravertebral block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- L - paravertebral block left: 30 woman above 18 years of age qualified for elective breast surgery on the left side of the body
  Interventions: Procedure: Paravertebral block (ropivacaine) left
- P - paravertebral block right: 30 woman above 18 years of age qualified for elective breast surgery on the right side of the body
  Interventions: Procedure: Paravertebral block (ropivacaine) right

INTERVENTIONS:
Procedure: Paravertebral block (ropivacaine) left — Paravertebral block at the level of 3rd thoracic intervertebral space on the left side. 0.5% Ropivacaine 0.3 ml·kg-1, not exceeding 30 ml, based on ideal body weight in obese patients
  Groups: L - paravertebral block left
Procedure: Paravertebral block (ropivacaine) right — Paravertebral block at the level of 3rd thoracic intervertebral space on the right side. 0.5% Ropivacaine 0.3 ml·kg-1, not exceeding 30 ml, based on ideal body weight in obese patients
  Groups: P - paravertebral block right

SUMMARY:
Aim of the study is to determine the presence and direction of electrocardiographical changes of cardiac repolarization after thoracic paravertebral block, depending on block laterality.

Injection of local anaesthetic into paravertebral space (paravertebral block, PVB) temporarily impairs transmission in nerve fibers in proximity of the deposition site. In case of PVB covering the rami of upper thoracic spinal nerves, among the others thoracic sympathetic cardiac nerves are blocked, possibly affecting action potential time of heart, especially the repolarization, and the related electrocardiographic phenomena.

The risk of life-threatening polymorphic ventricular tachycardia (torsade des pointes, TdP) is associated with certain electrocardiographical symptoms, like QT interval prolongation and increased transmural repolarization dispersion (TDR). Determining the presence and direction of cardiac repolarization changes after a thoracic PVB will allow to conclude about its impact on TdP risk: protective or, contrary, arrhythmogenic.

DETAILED DESCRIPTION:
After obtaining written informed consent, 60 women above 18 years of age scheduled to elective breast surgery in combined regional and general anaesthesia will be enrolled to study, divided in two groups depending of the side of operation. Participants will undergo the ultrasound-guided paravertebral block with single injection of 0.5% ropivacaine (0.3 ml·kg-1, not exceeding 30 ml, based on ideal body weight in obese patients) without adjuvants. Before injection (T0) and after confirmation of sufficient sensory block area covering 1st to 4th thoracic dermatomes (T1), 12-lead electrocardiogram (ECG) will be recorded using a Holter device. First examination of sensory block distribution will be performed 6 minutes after injection, with subsequent examinations if needed - every minute up to 15 minutes. No sedative premedication, general anaesthesia induction or additional medications (except of neutral saline maintaining intravenous access) will be administered until completions of ECG recording. Both T0 and T1 electrocardiogram will be preceded by rest in supine position for at least 5 minutes, without any medical procedures other than monitoring. Cases with baseline QT or corrected QT longer than 440 milliseconds (ms) will be excluded from study.

The QT interval and TDR (measured as time in milliseconds between ECG T wave peak [Tpeak] and end [Tend]) values obtained from baseline and post-blockade electrocardiograms will be statistically analyzed and compared between study groups.

The minimum sample size was calculated as 26 cases per study group, assuming a change in corrected QT of 20 milliseconds from the baseline value, with a significance level of p=0.05 and a test power of 0.9. Sample size was expanded to 30 cases per group, due to anticipated exclusions at the stage of intervention or data analysis.

ELIGIBILITY:
Inclusion Criteria:

* woman above 18 years of age, legally able of giving informed consent
* participants previously qualified for elective breast surgery due to neoplasm, with or without axillary node dissection
* physical status corresponding to class I or II in American Society of Anaesthesiologist classification

Exclusion Criteria:

* lack of consent to participation or to regional anaesthesia for planned surgery
* bilateral operation planned
* symptomatic circulatory disease at the time of qualification, artificial heart pacemaker presence, positive history of arrythmia
* allergy to amide local anaesthetics
* use of medications with "known" or "possible" potential of QT prolongation, according to Arizona Center for Education and Research on Therapeutics [AZCERT] Inc. list, in 5 days preceding the intervention
* severe deformation of thoracic spine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women above 18 years of age, without severe systemic comorbidities, patients of University Clinical Centre of Medical University of Gdańsk qualified for elective breast surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
QT interval | during procedure (6 minutes (prolonged until sufficient block distribution is achieved up to 15 minutes))
  difference in milliseconds of QT interval between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]
Corrected QT interval | during procedure (6 minutes (prolonged until sufficient block distribution is achieved up to 15 minutes))
  difference in milliseconds of QT interval corrected [according to Bazett, Framingham, Fredericia formulas] between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]
Tpeak-Tend | during procedure (6 minutes (prolonged until sufficient block distribution is achieved up to 15 minutes))
  difference in milliseconds of Tpeak-Tend time between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]

CONTACTS AND LOCATIONS:
Overall Officials: Radosław Owczuk, MD, PhD, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdańsk - Departament of Anesthesiology and Intensive Care, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided